CLINICAL TRIAL: NCT07021235
Title: Pilot Observational Cohort Study to Validate the Aiinane Preoperative and Preanesthesia Risk Assessment Tool in Real-world Conditions: Proof of Concept.
Brief Title: Proof of Concept of the Aiinane Preoperative Risk Assessment Tool.
Acronym: aiinane-24-1
Status: Completed | Type: Observational
Sponsor: Ancor Serrano (Other)
Collaborators: Hospital Universitari de Bellvitge (Other); Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Sponsor-Investigator, Ancor Serrano, MD, PhD,. Principal Investigator, Senior Consultant in Anesthesiology., Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Other Study IDs: ICPS033/24
Record Dates: First submitted 2025-05-28; First posted 2025-06-13 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Breast Neoplasms; Surgery Scheduled; Surgery Related Complications Rate; Preanesthetic Medication; Preoperative Patients; Preoperative Planning; Risk Assesment
Keywords: pre-anesthetic assessment; perioperative risk; artificial intelligence; Robotic Process Automation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer surgery: Adult patients diagnosed with breast cancer that require surgery as part of their treatment plan and have planed surgery in the following weeks.

SUMMARY:
BACKGROUND: Each year, over 13,000 patients in Catalonia and more than 4 million worldwide experience last-minute surgery cancellations (LMC) due to preoperative inefficiencies. As anaesthesia services struggle to meet surgical demands, thorough preoperative evaluations become challenging. Current resource-intensive pre-anaesthetic assessments are undermined by high demand, causing inefficiency. However, proper assessment identifies that most patients (>70%) are low-risk and ensures high-risk patients are adequately prepared by analyzing risk profiles, health status, medical history, treatment, and lab results.

RATIONALE: Previous attempts to improve preoperative risk assessment have mainly relied on self-administered questionnaires to detect at-risk patients. The investigators have identified a care model that enhances quality by adding value to preoperative risk assessment. By combining anaesthesiology expertise with AI techniques, the investigators developed an automated digital environment to detect risks, optimize visits, avoid cancellations, and reduce postoperative complications. This system uses parameterized medical knowledge to verify responses and objectively assess patient risk by integrating multiple data sources.

The investigators have developed a Class IIa active diagnostic and monitoring product, a Medical Device Software (MDSW, EMDN V92), to support clinical decision-making in an automated digital preoperative environment. It helps assess patients and flags low-risk from medium/high-risk individuals, reporting personalized needs to the medical team. The software was developed exclusively by independent researchers from Bellvitge University Hospital and the Bellvitge Biomedical Research Institute (IDIBELL).

HYPOTHESIS: The tool has been tested successfully on fictitious patients in controlled preclinical scenarios. The aim now is a proof-of-concept study to verify its performance with real patients in uncontrolled, real-world settings.

This is a Clinical Performance Research Study, aligned with MDSW Clinical Evaluation Guidelines (MDR, MDCG 2020-1) for (EU) 2017/745, and authorized by the Spanish Agency of Medicines and Medical Devices (AEMPS) and the local Ethics Committee.

MAIN OBJECTIVE: The clinical trial aims to verify that the software (aiinane), supporting preanesthetic assessment and preoperative risk estimation, is fit for its intended purpose and performs as expected under normal conditions of use.

This is an observational, non-interventional, single-center, prospective, longitudinal adult cohort study. The target population is any adult (>18 years) of any gender undergoing breast cancer surgery.

DETAILED DESCRIPTION:
The aiinane software has been developed by IDIBELL and HUB research staff. It is a software medical device (MDSW) with the intention of obtaining the CE marking under the modality 'class IIa active product'. The intention of this study is to take the first step towards obtaining the marking, as established by EU Regulation 2017 / 745.

The tool is in the preliminary development phase. An alpha version has been developed and executed within the hospital servers, in a simulated pre-production environment, with fictitious patients provided by the HUB.

Subsequently, a Beta version has been developed within the HUB servers, which has also been tested on simulated patients in the fictitious pre-production environment. The Beta phase is currently pending to be executed within the Hospital App 'ElMeuHUB', once it has been approved by the CEIm and the AEMPS to be tested in the real environment with real patients.

Intended purpose The aiinane tool is a computer programme designed to create a report where all the information collected and collated from different sources of information is shown in an aggregated manner. This report will include the results of applying the data collected to different risk scales/calculators already published in the scientific literature, preoperative risk assessment scales to assist the anaesthesiologist in decision making during the preoperative process.

It is expected that the aiinane software programme will be able to generate a final document for the healthcare professional with information on a patient, where a preoperative risk level is indicated and segmented, in order to support the healthcare professional (anaesthesiologist) in a pre-anaesthesia assessment.

Normal conditions of use:

The first condition of use is the one carried out by the patient. The patient must be able to answer a personalised health questionnaire and complete it by interacting via a WebApp hosted within the 'ElMeuHUB' App, the HUB's official App. To access the questionnaire, the patient must have installed ElMeuHUB and have enabled personal and unique access to his/her private area within the application. This is the only way to access the AIINANE questionnaire.

The second condition of use is that of the researcher (in the future, the clinical care staff). They must be able to access the back-office and obtain the complete report for an individual patient with the information provided by the tool. The back-office is only available within the hospital servers and during the present study only to the hospital researchers.

Manufacturer. The software is designed, written, developed and compiled by members of the 'Perioperative Pathophysiology and Pain' research group, within the Neurosciences area of IDIBELL - Bellvitge Biomedical Research Institute - and the Anaesthesiology, Resuscitation and Pain Treatment Service of the Bellvitge University Hospital.

The team responsible for the project is made up of both anaesthesiologists with extensive experience in their field of work, and computer engineers. Thus, the different profiles of the team complement each other in different fields of knowledge to create a multidisciplinary team. This allows them to have the necessary experience and knowledge to be able to carry out the development and purpose of the tool, as well as its implementation for the proof of concept.

According to the laws 1/1996 of 12 April, 1/2015 and 611/2023 of 11 July, the owner of the programme is the employer of the team. In this case the Institut Català de la Salut (ICS), as the public company responsible for the HUB, with registered office at Gran via de les Corts Catalanes, 587, Barcelona, Spain, with CP: 08007 and NIF Q5855029D; and the Institut d'Investigació Biomèdica de Bellvitge (IDIBELL), as a research foundation related to the HUB, with registered office at Gran via de L'Hospitalet 199-203, 2ª planta, de L'Hospitalet de Llobrgat, 08908 (Barcelona - SPAIN) and NIF G58863317.

Traceability.

Traceability has 3 components:

1. The traceability of the aiinane tool itself. That which a competent authority may require to check how the product has been developed and which can be explained and followed by someone with knowledge in the field. The tools and programmes that have been used to develop the aiinane programme are described in an internal document, kept in the same place as the programme, to avoid loss of intellectual property rights. At the time of registration of these rights and during the CE marking procedure, it will be attached with the required documentation. In the meantime, it is available for audits or inspections.

   Both the software and the databases for its implementation are integrated within the HUB's own servers. The hospital servers have a record of who has executed calls to the server and can control access and review past actions. In addition, the aiinane programme creates records of the actions taken by the programme, including who initiated the action, who performed the action and at what time it was performed.
2. Traceability of the CRD-e Access to the CRD-e will have traceability of who accesses it, when they access it and the changes they make, once they have been saved and signed.
3. Traceability of the data collected by the aiinane tool. The data that the tool collects and then presents to the doctor will have a record of the date on which the data is collected, as well as the date on which the report is generated. The tool also collects date traceability internally to be able to check if there is new data to be submitted, and/or if the pre-operative is being delayed and the surgery date is approaching.

Contact with the human body. A risk assessment tool is being evaluated based on data collected from medical records and a questionnaire filled in by patients using their mobile devices. There is no contact with the human body beyond the contact each patient has with her mobile device as for any other daily task.

Risk assessment A separate document has been developed with a risk analysis, risk mitigation and contingency plans. It can be found in the Annex to the protocol and has been supervised and approved by both the competent authority and the research ethics committee.

e-CRF: Once the patient has signed the Informed Consent, the investigator will enter data corresponding to visit 1 in the CRD-e. In the EHR, he/she will record the subject number in the CRD-e and then save this information in the separate document for this purpose.

Subsequently, THEY WILL NOT HAVE ACCESS TO THE TOOL RESULT UNTIL VISIT 2, which will be 14 ±3 days after the patient has undergone surgery. In other words, the patient's profile in the aiinane programme will not be seen by the staff until after the surgery has been performed.

Screening Failure Currently, as it is not CE marked, the device being tested in this clinical investigation is designed, for safety reasons, to be used solely and exclusively within the hospital's IT systems, i.e. through the personal area within the Hospital's native App that must be downloaded from official stores (Google Play or Apple Store).

Therefore, there are patients who meet all the inclusion criteria, do not meet any of the exclusion criteria and wish to participate, BUT, after signing the informed consent, they have problems downloading the official ElMeuHUB Hospital App, either because their usual device is a company device and downloads are restricted, or because the contact details provided by the hospital are not the same as those they normally use and enter in the personal area of the App.

These patients cannot continue with the study process for reasons beyond the control of the MDSW device itself. Therefore, they will be assigned as a screening failure.

Patients who wish to participate initially, but do not finish the preoperative assessment before the surgery will be considered as they have withdrawn their consent, being screening failure too.

Withdrawal of subjects from the study No withdrawal of subjects from the study is foreseen a priori, as this is a proof-of-concept study, with an interval between inclusion and preoperative assessment. However, patients may not complete the preoperative assessment questionnaire. Encountering subjects who do not complete the questionnaire is itself part of the proof of concept. It is part of the stress scenario that the aiinane application will be subjected to, not having all sources of information, as well as not being able to obtain data from the electronic medical record because the patient comes from another hospital system.

Care of patients after the end of the study After the end of the clinical trial, participating patients will continue to be followed by their surgeons and the respective oncology team. They will continue with the tests and treatments prescribed to them, in accordance with standard clinical practice.

Statistical considerations.

1. Sample size determinations As this was an exploratory study, the sample size calculation was not based on hypothesis testing. The sample size was defined on the basis of the total number of patients meeting the inclusion criteria during the study period.

   In one year, about 700 breast surgery procedures are performed at Bellvitge University Hospital. An acceptance rate (consent to participate) of 50% is estimated. In an approximate duration of 2 months it is expected to be able to recruit 30 patients.
2. Statistical analysis Because this is a pilot study with a very small number of patients, it is not intended to achieve statistical significance, but descriptive significance. However, whenever possible, various statistical tests will be performed to assess the independence or relationship between the categorised variables, such as the chi-square test (χ²) and Fisher's exact test.

An exploratory analysis will be performed on the clinical significance of the data especially the alerts (if and when they appear) and the risk calculators, as well as their correlation with the ASA classification system, or their superiority (in level of detail and/or segmentation).

Monitoring This trial will be supervised by the monitor in accordance with ICH GCP principles and Regulation (EU) 2017/745. This is to ensure that the safety and rights of participants are protected and that the trial is conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements.

During monitoring, any data inconsistencies detected during source data verification, safety review, or data management review will be investigated. A single follow-up visit will be conducted one month after the first patient is enrolled, and a final visit, given the short duration of the study. During these visits, the monitor will review the following information:

* Verify the latest version of the protocol and other approved documents, if any amendments have been made.
* Informed consent forms and their procedures.
* 100% source document verification
* Significant protocol deviations
* Personnel changes
* Definitions of adverse events and serious adverse events, reporting procedures, and contact information
* Completion, error correction, and maintenance of the CRF
* Source documentation requirements
* Device accountability requirements
* Principal investigator qualifications and resources
* Site personnel, facilities, storage, and equipment are adequate to conduct the research safely and appropriately
* Suitability and accessibility of the participant population
* Access to source documentation
* Any other issues deemed important to the conduct of the study

In summary, the monitor will play an important role in the successful conduct of the study. Anyone with direct access to the data (Regulatory Authorities, Trial Monitors, and auditors) will take every precaution to maintain the confidentiality of patient identities.

It is the responsibility of the Investigator to obtain informed consent from the patient in the study, and the Trial Monitor to verify that each patient has given written consent to allow this direct access.

All parties involved in the study agree to direct access to source data and study-related documents and reports, for monitoring and auditing by the Sponsor, and for inspection by the Regulatory Authorities.

Audit. An audit consists of the systematic and independent examination of the study-related activities and documents to determine whether they were performed, and whether the data were recorded, analyzed, and reported, in accordance with the protocol, the Sponsor's Standard Operating Procedures, good clinical practices (GCP), and applicable regulations.

The Investigator will allow a person designated by the Sponsor to audit the facilities and documentation at agreed times. The auditors must be independent of the clinical trial and its conduct.

Inspection. An inspection is the act by which the Regulatory Authorities conduct an official review of documents, facilities, records, and other resources they deem relevant to the clinical trial and that may be located at the Study Center or the Sponsor's facilities. The Investigator must cooperate with any inspection.

Protocol Amendments Any changes to the protocol during the study will be recorded as amendments along with a new version of the protocol. These will be signed by the Sponsor and the Principal Investigator.

Depending on the content of the amendment and local legal requirements, the amendment will be submitted for approval by the corresponding REC and the Spanish Medicines Agency (EU Regulation 2017/745).

No significant deviations or changes to the protocol will be made without prior review and approval by the REC and the relevant Competent Authority, except when necessary to eliminate an imminent risk to patients, or when the change(s) involve only logistical or administrative aspects of the clinical trial. Prospective approval of protocol deviations from the recruitment and enrollment criteria, also known as protocol waivers, is not permitted.

If a modification substantially affects the clinical trial design, potential patient risks, or patient treatment, the Patient Information Sheet will be revised and submitted to the appropriate IRB and Competent Authorities for review and approval.

When a patient undergoing clinical trial procedures is affected by a modification, the patient's Informed Consent will be requested again, using the new version of the Patient Information Sheet. If the enrollment period has not been completed, the new version of the Patient Information Sheet will be used to obtain consent from patients who continue to be enrolled in the study.

Protocol deviations (PDs) are unplanned perversions of the research protocol or noncompliance with it. PDs will be identified and documented during the course of the research. PDs are classified according to their impact on subject well-being or data quality. The sponsor or its representative is responsible for promptly and regularly submitting PD reports to the relevant regulatory authorities (AEMPS and IRB), in accordance with local regulatory requirements.

Serious breaches are described as violations of GCP or PD that have a significant impact on the safety and rights of a patient, or on the reliability and robustness of the data generated by the clinical investigation (Regulation (EU) 2017/745). During the course of the investigation, serious breaches will be identified and documented and immediately reported to the sponsor. The sponsor is responsible for reporting the serious breach to the competent authority within 7 calendar days of becoming aware of it.

Limitations of the design, data source, and analysis methods. This study is based on the prospective observation of a cohort of patients treated at Bellvitge University Hospital (tertiary care hospital) for a limited period from its inception (inclusion period), subject to authorization from the competent authorities. Therefore, the main expected biases would be those characteristic of cohort studies.

* Observation bias. When attempting to extract, link, and structure data, observation bias may arise from the tool itself. The researcher only needs to assess the tool's performance (whether it extracts data and produces a report with that data). Observation bias is limited to the source (electronic medical records) having incorrect data.
* Presence of confounding factors. Since this is primarily a descriptive study, it is considered that this bias will not influence the final results of the study.

Due to its design, the medical record may not contain the information intended for this study. However, this is a possibility that can occur in real-life practice, and one of the objectives of this study is to verify the proper functioning of the aiinane tool when relevant information is missing (i.e., its ability to generate an alert during the preoperative assessment regarding the absence of such relevant information).

Ethical Aspects/Protection of Participating Subjects

1. Ethical Considerations This study will be conducted in accordance with the basic ethical principles contained in the Declaration of Helsinki (Revision of the 64th General Assembly, Fortaleza, Brazil, October 2013), GCP, and applicable regulations. GCP is a standard for clinical trials (design, conduct, development, monitoring, auditing, recording, analysis, and communication) that ensures that the data and results reported are credible and accurate, and that the rights, integrity, and confidentiality of patients are protected.

   The protocol will be reviewed by the Research Ethics Committee of Bellvitge University Hospital. The study may only begin once the IEC has given its signed and dated approval of the protocol, as well as the Patient Information Sheet and Informed Consent forms.

   The researchers' participation in this study is free, voluntary, and unpaid.

   The investigator is responsible for ensuring that the clinical trial is conducted in accordance with the protocol, the guidelines established by the International Conference on Harmonization (ICH) on GCP, and local legal requirements.

   Each person involved in the conduct of the study must be qualified by education, training, and experience to perform their specific duties.

   Neither the investigators nor the study staff will coerce or pressure patients to participate or continue in the study. The investigator may not include themselves, their family members, or members of their clinical team or their family members in the study.
2. Safety 2.1) Benefit-risk assessment of research subjects. This study is based on the collection of information from the patient's medical history and a patient questionnaire. The results obtained from this information will not influence clinical practice. This will be routine and independent of the information collected and the report generated by the aiinane tool. Therefore, no risk to the research subjects is anticipated.

2.2) Adverse Event Management. Since there is no interference with routine clinical practice, no adverse events related to the tool are expected. However, since data is collected from the medical record, events may be identified due to any medication the patient is taking or prescribed during the treatment.

2.3) Pregnancy Pregnancy is an exclusion criterion. If a pregnancy occurs during the study, the investigator will notify the sponsor or whoever assumes the sponsor's delegated duties within 24 hours of becoming aware of the pregnancy, and the patient will be withdrawn from the study. If the pregnancy outcome meets the criteria for an AEG or if the newborn presents a serious event, the procedures described for AEG notification will be followed.

Notification will be made using the specific pregnancy notification form, which will be sent by FAX or email to the same contact who will receive AAG notifications.

Although this research study does not affect clinical practice, with the healthcare system operating in parallel with healthcare activity without intervention on the patient, EU Regulation 2017/745 and the applicable law in the Spanish State, Royal Decree 192/2023, of March 21, which regulates medical devices, both require the detailed monitoring plan for Adverse Events, even if they are not anticipated.

Therefore, adverse effects will be monitored and followed in accordance with the legal requirements requested by the authorities in the aforementioned regulations.

Considerations Regarding Subject Information and Informed Consent Before performing any study-related procedure, the researcher will be responsible for providing each patient (or legal representative, if applicable) with the Patient Information Sheet specifically prepared and approved for the study, which the patient must read.

Understandable language will be used to inform them about the research treatments, the objectives of the study, and the advantages and disadvantages of participating in the study.

Patients will be given sufficient time to consider their participation, and any questions they may have will be answered.

The researcher will inform patients that their participation in the study is voluntary and that they are free to voluntarily withdraw from the study at any time and for any reason. Their decisions will not affect the treatment they receive from their physicians, and they will not incur any penalties or loss of benefits to which they are otherwise entitled. In any case, the Researcher should try to rule out an adverse event as the reason for voluntary withdrawal.

The researcher will be responsible for obtaining written informed consent from each participating patient before proceeding with any medical procedure specific to the study. Agreement to participate in the clinical trial will be expressed by signing and dating the Informed Consent document specifically prepared and approved for the study. The researcher who led the Informed Consent process must also sign and date the Informed Consent document.

The Informed Consent document will be signed in duplicate; one original copy will be given to the patient or their legal representative, and the other original copy will be retained by the researcher.

If new information arises during the course of the study that could affect the informed consent process, the Patient Information Sheet will be revised. Before it can be used, the revised version will be submitted for approval by the Ethics Committee.

The patient will be informed as soon as possible if new information becomes available that could affect the patient's decision to continue in the study. The communication of this information must be recorded. The patient, or his or her legal representative, will receive a copy of any updates to the Informed Consent or any other relevant written information.

Interference with the physician's prescribing habits. None. This is an observational study to verify that, under normal conditions of use, the study tool is suitable for its stated purposes and performs as intended.

There is no interference with clinical practice. The results of the tool will not be used for clinical decision-making.

The results presented by the aiinane program will be evaluated by the research team

Specific Clinical Trial Insurance As this is a study involving a medical device (MD MDSW), the applicable legislation in Spain for clinical research involving medical devices is Royal Decree 192/2023, of March 21, regulating medical devices. Article 32 of this Decree regulates aspects related to compensation for damages in the field of clinical research involving medical devices.

Although this is an observational, non-interventional study, and therefore lower risk than a "low-intervention clinical trial," a civil liability insurance policy must still be in place, in accordance with Royal Decree 192/2023, of March 21, regulating medical devices.

Therefore, this policy has been taken out.

Funding. This study is an independent study. It is partially funded by the researchers' own resources. To conduct part of the study, the team is seeking funding from various sources, such as a competitive grant from a public administration or donations from private foundations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years) of both sexes. Although breast neoplasia is a pathology with high prevalence in the female biological gender, we do not rule out recruiting patients of male biological gender.
* Who have been indicated for breast surgery to resolve breast cancer pathology.
* Who will undergo a pre-anesthetic evaluation during the inclusion period..
* Subjects must understand the nature of the study procedures and provide written informed consent prior to any study-related procedures.

Exclusion Criteria:

* Surgery scheduled for <7 days from enrollment
* Inability to participate in the study, in the opinion of the investigator, due to, for example, severe brain damage, language barrier, dementia, or other clinically significant or unstable conditions.
* Subject's participation in any other clinical study.
* Subjects dependent (as employee or relative) of the promoter or researcher.
* Subjects placed in an institution by virtue of an order issued by either judicial or administrative authorities.
* Limited legal capacity or incapacity.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target population: patients who will undergo preanesthetic evaluation at Bellvitge University Hospital for breast cancer surgery.
  An internal analysis performed on all types of surgical procedures in 2019 (2020 to 2022 skewed due to the COVID-19 pandemic) identified 4 types of surgery with 80% of patients categorized preoperatively as ASA I-II (low risk). From those, breast cancer surgery was the only one with a short intervention period between diagnosis, surgical indication and surgery.
  Patients who will undergo breast cancer surgery go through multiple visits, tests and treatments between diagnosis and surgery. Sparing them visits generates a high impact on their emotional state.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
The aiinane tool is able to create a final report/document with the clinical information required for preoperative assessment | From enrollment to 2 weeks after surgery has been performed.
  The present clinical trial aims to verify that the software (hereinafter aiinane) for the support of pre-anesthetic assessment in the estimation of preoperative risk, is adequate for its established purposes and offers the expected performance under normal conditions of use.
  Therefore the outcome measure is the total number of complete anesthesia reports generated.

SECONDARY OUTCOMES:
Patient Satisfaction | From enrollment to 2 weeks after surgery
  Evaluate patient satisfaction with the use of the digital tool for preoperative evaluation.
  This will be evaluated with 2 questions. First question. Patient satisfaction in dichotomous yes/no answer. Second question. Rate of satisfaction in a 5 point Likert score, with 1 being totally dissatisfied and 5 being totally satisfied.
Clinical usefulness | From enrollment to 2 weeks after surgery
  Evaluate whether the completed report is useful to the anesthesia service.
  This will be evaluated with 2 questions. First question. Is the resport usefurl in dichotomous yes/no answer. Second question. Rate ofusefulness in a 5 point Likert score, with 1 being completely useless and 5 being completely useful.
clinical significance | From enrollment to 2 weeks after surgery
  Evaluate whether the overall risk level report has clinical significance.
  This will be evaluated with 2 questions. First question. Is the resport usefurl in dichotomous yes/no answer.
  Second question. Rate of significance in a 5 point Likert score, with 1 being totally insignificant and 5 being completely significant.
usefulness of risk stratification | From enrollment to 2 weeks after surgery
  Evaluate whether the different risk stratifications presented by aiinane are useful.
  This will be evaluated with 2 questions. First question. Is the resport usefurl in dichotomous yes/no answer. Second question. Rate ofusefulness in a 5 point Likert score, with 1 being completely useless and 5 being completely useful.

CONTACTS AND LOCATIONS:
Overall Officials: Ancor Serrano Afonso, MD, PhD, Principal Investigator — Bellvitge University Hospital
Locations (1):
- Bellvitge University Hospital. ,, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
A decision has not yet been made as to which data collected in the Case Report Form are subject to further intellectual property rights protection. A rights protection analysis must be performed before the IPD dissemination plan can be made.

REFERENCES:
- [Background] Al Talalwah N, McIltrot KH. Cancellation of Surgeries: Integrative Review. J Perianesth Nurs. 2019 Feb;34(1):86-96. doi: 10.1016/j.jopan.2017.09.012. Epub 2018 Apr 17. PMID 29678319
- [Background] Glazener C, Boachie C, Buckley B, Cochran C, Dorey G, Grant A, Hagen S, Kilonzo M, McDonald A, McPherson G, Moore K, N'Dow J, Norrie J, Ramsay C, Vale L. Conservative treatment for urinary incontinence in Men After Prostate Surgery (MAPS): two parallel randomised controlled trials. Health Technol Assess. 2011 Jun;15(24):1-290, iii-iv. doi: 10.3310/hta15240. PMID 21640056
- [Background] Finegan BA, Rashiq S, McAlister FA, O'Connor P. Selective ordering of preoperative investigations by anesthesiologists reduces the number and cost of tests. Can J Anaesth. 2005 Jun-Jul;52(6):575-80. doi: 10.1007/BF03015765. PMID 15983141
- [Background] Rogers G. Using Telemedicine for Pediatric Preanesthesia Evaluation: A Pilot Project. J Perianesth Nurs. 2020 Feb;35(1):3-6. doi: 10.1016/j.jopan.2019.07.001. Epub 2019 Sep 11. PMID 31521494
- [Background] Kramer S, Lau A, Kramer M, Wendler OG, Muller-Lobeck L, Scheding C, Klarhofer M, Schaffartzik W, Neumann T, Krampe H, Spies C. [Web-based for preanesthesia evaluation record: a structured, evidence-based patient interview to assess the anesthesiological risk profile]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2011 Oct;46(10):694-8. doi: 10.1055/s-0031-1291948. Epub 2011 Oct 21. German. PMID 22020575
- [Background] Schoen DC, Prater K. Role of Telehealth in Pre-anesthetic Evaluations. AANA J. 2019 Feb;87(1):43-49. PMID 31587743
- [Background] Gonzalez-Arevalo A, Gomez-Arnau JI, delaCruz FJ, Marzal JM, Ramirez S, Corral EM, Garcia-del-Valle S. Causes for cancellation of elective surgical procedures in a Spanish general hospital. Anaesthesia. 2009 May;64(5):487-93. doi: 10.1111/j.1365-2044.2008.05852.x. PMID 19413817
- [Background] Seim AR, Fagerhaug T, Ryen SM, Curran P, Saether OD, Myhre HO, Sandberg WS. Causes of cancellations on the day of surgery at two major university hospitals. Surg Innov. 2009 Jun;16(2):173-80. doi: 10.1177/1553350609335035. Epub 2009 May 21. PMID 19460816
- [Background] Connor CW. Artificial Intelligence and Machine Learning in Anesthesiology. Anesthesiology. 2019 Dec;131(6):1346-1359. doi: 10.1097/ALN.0000000000002694. PMID 30973516
- [Background] Vetter TR, Boudreaux AM, Ponce BA, Barman J, Crump SJ. Development of a Preoperative Patient Clearance and Consultation Screening Questionnaire. Anesth Analg. 2016 Dec;123(6):1453-1457. doi: 10.1213/ANE.0000000000001532. PMID 27529323
- [Background] Manso M, Schmelz J, Aloia T. ERAS-Anticipated outcomes and realistic goals. J Surg Oncol. 2017 Oct;116(5):570-577. doi: 10.1002/jso.24791. Epub 2017 Sep 5. PMID 28873504
- [Background] Committee on Standards and Practice Parameters; Apfelbaum JL, Connis RT, Nickinovich DG; American Society of Anesthesiologists Task Force on Preanesthesia Evaluation; Pasternak LR, Arens JF, Caplan RA, Connis RT, Fleisher LA, Flowerdew R, Gold BS, Mayhew JF, Nickinovich DG, Rice LJ, Roizen MF, Twersky RS. Practice advisory for preanesthesia evaluation: an updated report by the American Society of Anesthesiologists Task Force on Preanesthesia Evaluation. Anesthesiology. 2012 Mar;116(3):522-38. doi: 10.1097/ALN.0b013e31823c1067. No abstract available. PMID 22273990
- [Background] Sabate S, Gomar C, Canet J, Castillo J, Villalonga A; Grupo ANESCAT. [Survey of anesthetic techniques used in Catalonia: results of the analysis of 23,136 anesthesias (2003 ANESCAT study)]. Rev Esp Anestesiol Reanim. 2008 Mar;55(3):151-9. doi: 10.1016/s0034-9356(08)70533-4. Spanish. PMID 18401989
- See also: Population statistics published by the Statistical Agency of the Generalitat de Catalunya (g — https://www.idescat.cat/indicadors/?id=basics&n=10328&lang=en
- See also: Institut Catalan de la Salut's 2018 activity report. — https://scientiasalut.gencat.cat/bitstream/handle/11351/4555/servei_catala_sa%20lut_memoria_2018.pdf?sequence=4&isAllowed=y